CLINICAL TRIAL: NCT03912077
Title: War and Immigration: Implementing Psychosocial Interventions to Syrian Refugee Women Who Are Exposed to Psychological Trauma
Brief Title: Implementing Psychosocial Interventions to Syrian Refugee Women Who Are Exposed to Psychological Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sehir University (Other)
Responsible Party: Principal Investigator, Halime Sevde Eskici, Principal Investigator, Istanbul Sehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/2018No:1
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Psychological Distress; Psychological Trauma
Keywords: Refugees; Psychological distress; Psychological trauma; Anxiety; CA-CBT; Depression; Post-traumatic stress disorder; Intervention; Turkey; Migration
MeSH Terms: conditions — Psychological Trauma; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: It is a randomized, parallel-group trial that enroll Syrian refugee women with psychological distress, according to the Hopkins Symptom Checklist - 25 (HSCL-25) who will be randomly assigned to the Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) intervention or to treatment as usual (TAU).
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blind to the study conditions; while participants and facilitators will be aware of the study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally Adapted Cognitive Behavioural Therapy (Experimental): Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) is an evidence-based psychological intervention manual developed by Devon Hinton, MD from Harvard University and Baland Jalal from University of Cambridge. It is a group therapy protocol that consists of 7 sessions.
  It is a brief, feasible and culturally sensitive intervention that has a transdiagnostical approach. Detailed information about Syrian culture, idioms of stress, cultural differences, and psychological problems that Syrian refugee women have been facing and their needs, expectations and sensitivities are considered in the adaptation process. Examples, cultural metaphors and imageries that take part in the manual are adapted according to Syrian culture.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioural Therapy
- Treatment as Usual (No Intervention): Control arm participants will receive routine social support and/or care according to ordinary practice of the non-governmental organization (treatment as usual). Also, they will receive baseline and post assessments according to the study schedule.

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioural Therapy — 7-session psychosocial intervention
  Arms: Culturally Adapted Cognitive Behavioural Therapy

SUMMARY:
This study assesses severity of trauma, depression and anxiety symptoms of Syrian women under temporary protection who reside in Istanbul and types of exposed trauma that they have experienced. This study also evaluates the effectiveness of the Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) in Syrian women under temporary protection who are with psychological distress in Turkey. Half of participants will receive Culturally Adapted Cognitive Behavioural Therapy (CA-CBT), while the other half will receive treatment as usual.

DETAILED DESCRIPTION:
Background: Due to the ongoing conflict in Syria, Syrian people have faced with various atrocities. Many of them were displaced from their home, causing them to experience difficulties during and after the immigration. Being exposed to such stressors makes refugees susceptible to psychological distress and put them at risk to develop psychological disorders such as post-traumatic stress disorder, anxiety disorders, depression and so on (Alpak et al., 2015).

Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) is an evidence-based psychological intervention manual developed by Devon Hinton, MD from Harvard University and Baland Jalal from University of Cambridge. It is a group therapy protocol that consists of 7 sessions. CA-CBT is a brief intervention that adopts a transdiagnostical approach and can be delivered by trained facilitators to people who are psychologically distressed. Several RCTs has been conducted to evaluate effectiveness of CA-CBT and demonstrated positive results. (Hinton et al., 2012).

Objectives: This study has two aims. First aim of the study is to assess severity of trauma, depression and anxiety symptoms and types of exposed trauma of Syrian refugee women who reside in Istanbul. Second aim of the study is to evaluate the effectiveness of the Culturally Adapted Cognitive Behavioural Therapy in Syrian refugee women with psychological distress resettled in Turkey, as compared with treatment as usual (TAU). The primary outcome is the decrease in psychological distress symptoms. Secondary outcomes are depression, anxiety and psychological trauma symptoms along with post-migration living difficulties and related distress symptoms.

Design: This is a parallel-group randomized controlled trial, therefore participants will have an equal probability (1:1) of being randomly allocated to the CA-CBT intervention or the TAU.

Methodology: Screening will be conducted before randomization. Syrian refugee women who score 1.75 or above (≥ 1.75) at the Hopkins Symptom Checklist - 25 (HSCL-25) will enter the study. After randomization they will receive the 7- session CA-CBT or the TAU. The CA-CBT intervention phase will last 7 weeks (1 session per week). After intervention, post-assessments will be performed.

Expected outcomes: The expected outcome is decrease in the depression, anxiety and psychological trauma symptoms and general improvement in distress symptoms caused by post-migration living difficulties, in refugees in the CA-CBT intervention arm, as compared to TAU.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old and older
* Being a Syrian woman under temporary protection who resides in Istanbul
* Being able to speak and understand Arabic
* Having psychological distress symptoms, as shown by a score of 1.75 or more at the Hopkins Symptoms Checklist-25 (HSCL-25 ≥ 1.75 )

Exclusion Criteria:

* Imminent risk of suicide
* Severe mental disorder (psychotic disorders, substance dependence)
* Severe cognitive impairment (severe intellectual disability or dementia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Psychological distress symptoms | 1-week post-intervention
  Hopkins Symptoms Checklist - 25 (HSCL-25) measures psychological distress symptoms and has 25 items. Participants rate each item from 1 (not at all) to 4 (extremely). First 10 items measure anxiety symptoms, whereas the following 15 items measure depression symptoms. There are many studies, which demonstrate that the Arabic version of HSCL-25 is statistically reliable and valid (Kobeissi et al., 2011). HSCL-25 has been used in several intercultural studies (Aragona et al., 2013) and cut-off score has been assigned as 1.75 in many studies (Hasanović and Herenda, 2008). The current study will primarily look at the total score in which the lower values represent a better outcome.

SECONDARY OUTCOMES:
Psychological trauma symptoms | 1-week post-intervention
  Harvard Trauma Questionnaire (HTQ) assesses the traumatic events that one experienced during his/her lifetime (Part I of the questionnaire) and measures the severity of post-traumatic stress disorder symptoms (Part IV of the questionnaire) (Mollica et al., 2004). The first part of the HTQ consists of 43 traumatic events and participants are asked to answer whether they have experienced such traumatic event or not, by choosing 'Yes' or 'No'. The fourth part of the HTQ has 45 items and participants are asked to rate each item from 1 (not at all) to 4 (extremely).
Depression symptoms | 1-week post-intervention
  Beck Depression Inventory II (BDI-II) measures depression symptoms and has 21 items. The total score of BDI-II varies from 0 to 63 and higher scores indicate more severe depressive symptoms (Beck et al., 1996). The Arabic version of the BDI-II has been developed by Ghareeb (2000).
Distress symptoms related with post-migration events | 1-week post-intervention; 6-month and 12-month follow-ups
  Post-Migration Living Difficulties (PMLD) assesses adverse events that one experienced after migration and measures the distress level induced by such events. Participants are asked to evaluate their experiences regarding the problems they had in the last 12 months. PMLD has 17 items and participants are asked to rate each item from 0 (was not a problem/did not happen) to 4 (a very serious problem).

CONTACTS AND LOCATIONS:
Locations (1):
- Refugees and Asylum Seekers Assistance and Solidarity Association, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alpak G, Unal A, Bulbul F, Sagaltici E, Bez Y, Altindag A, Dalkilic A, Savas HA. Post-traumatic stress disorder among Syrian refugees in Turkey: a cross-sectional study. Int J Psychiatry Clin Pract. 2015 Mar;19(1):45-50. doi: 10.3109/13651501.2014.961930. Epub 2014 Oct 6. PMID 25195765
- [Background] Hinton DE, Rivera EI, Hofmann SG, Barlow DH, Otto MW. Adapting CBT for traumatized refugees and ethnic minority patients: examples from culturally adapted CBT (CA-CBT). Transcult Psychiatry. 2012 Apr;49(2):340-65. doi: 10.1177/1363461512441595. PMID 22508639
- [Background] Kobeissi L, Araya R, El Kak F, Ghantous Z, Khawaja M, Khoury B, Mahfoud Z, Nakkash R, Peters TJ, Ramia S, Zurayk H. The relaxation exercise and social support trial-resst: study protocol for a randomized community based trial. BMC Psychiatry. 2011 Aug 25;11:142. doi: 10.1186/1471-244X-11-142. PMID 21864414
- [Background] Aragona M, Pucci D, Mazzetti M, Maisano B, Geraci S. Traumatic events, post-migration living difficulties and post-traumatic symptoms in first generation immigrants: a primary care study. Ann Ist Super Sanita. 2013;49(2):169-75. doi: 10.4415/ANN_13_02_08. PMID 23771261
- [Background] Hasanovic M, Herenda S. Post traumatic stress disorder, depression and anxiety among family medicine residents after 1992-95 war in Bosnia and Herzegovina. Psychiatr Danub. 2008 Sep;20(3):277-85. PMID 18827753
- [Background] Ghareeb, A. G. Manual of the Arabic BDI-II. Cairo, Egypt: Angle Press. 2000.
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. Manual for Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation. 1996.
- [Background] Silove D, Sinnerbrink I, Field A, Manicavasagar V, Steel Z. Anxiety, depression and PTSD in asylum-seekers: assocations with pre-migration trauma and post-migration stressors. Br J Psychiatry. 1997 Apr;170:351-7. doi: 10.1192/bjp.170.4.351. PMID 9246254
- [Background] Shoeb M, Weinstein H, Mollica R. The Harvard trauma questionnaire: adapting a cross-cultural instrument for measuring torture, trauma and posttraumatic stress disorder in Iraqi refugees. Int J Soc Psychiatry. 2007 Sep;53(5):447-63. doi: 10.1177/0020764007078362. PMID 18018666
- [Background] Mollica, R. F., McDonald, L. S., Massagli, M. P., & Silove, D. Measuring trauma, measuring torture: instructions and guidance on the utilization of the Harvard Program in Refugee Trauma's Versions of the Hopkins Symptom Checklist-25 (HSCL-25) & The Harvard Trauma Questionnaire (HTQ). Harvard Program in Refugee Trauma. 2004.
- [Derived] Eskici HS, Hinton DE, Jalal B, Yurtbakan T, Acarturk C. Culturally adapted cognitive behavioral therapy for Syrian refugee women in Turkey: A randomized controlled trial. Psychol Trauma. 2023 Feb;15(2):189-198. doi: 10.1037/tra0001138. Epub 2021 Oct 7. PMID 34618479